CLINICAL TRIAL: NCT06791057
Title: Multi-site Trial of a Brief Behavioral Intervention for Dyspnea in Patients With Advanced Lung Cancer
Acronym: BREEZE+
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Johns Hopkins University (Other); University of Miami (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Temel, MD, co-Prinipal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24-657; R01CA292902 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Advanced Lung Cancer; Dyspnea
Keywords: Dyspnea; Breathlessness; Lung Cancer; Behavioral Intervention
MeSH Terms: conditions — Dyspnea; Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyspnea Intervention (Experimental): Patients will receive three nurse-delivered sessions that focus on: (1) psychoeducation about the relationship between dyspnea and the physiologic stress response, (2) behavioral techniques for managing acute episodes of breathlessness (i.e., pursed-lip breathing, postural positions, and fan therapy), and (3) skills for reducing physiologic stress and strengthening lung capacity (e.g., slow diaphragmatic breathing; mindful breathing). Patients will also receive a digital health app downloaded to their mobile phone to reinforce daily practice of the dyspnea management skills. Patients may receive any usual care for their dyspnea as deemed appropriate by their clinicians.
  Interventions: Behavioral: Dyspnea Intervention
- Enhanced Usual Care (Active Comparator): Patients will receive printed or electronic handouts regarding the common symptoms and side effects of lung cancer, including dyspnea, and recommendations for management from the American Cancer Society, with a link to their website of patient-education materials. Patients may receive any usual care for their dyspnea as deemed appropriate by their clinicians.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Dyspnea Intervention — Brief behavioral intervention for dyspnea management that includes three nurse-led sessions focused on psychoeducation, behavioral techniques for managing acute breathlessness, and relaxation training for reducing physiological stress as well as a digital health app to reinforce practice of breathing skills.
  Arms: Dyspnea Intervention
Behavioral: Enhanced Usual Care — Patients will receive educational materials on the management of symptoms of lung cancer and its treatment as well as any usual care for dyspnea deemed appropriate by the clinical team.
  Arms: Enhanced Usual Care

SUMMARY:
Dyspnea, or breathlessness, is one of the most common and distressing symptoms experienced by patients with advanced lung cancer. The purpose of this multi-site trial is to test the effectiveness of a dyspnea intervention (called BREEZE+) that includes three brief nurse-delivered sessions and access to a digital health app that teaches and reinforces patients' use of skills for managing and coping with this highly debilitating symptom. This study will lay the groundwork for a follow-up pragmatic implementation trial integrating BREEZE+ into usual oncology care for patients with advanced lung cancer experiencing dyspnea.

DETAILED DESCRIPTION:
The goal of this study is to improve dyspnea, one of the most common and debilitating symptoms experienced by patients with advanced lung cancer. Despite improvements in survival from novel targeted therapy and immunotherapy for patients with advanced lung cancer, the proportion of patients experiencing dyspnea (i.e., difficulty breathing) has not decreased. In fact, recent data show that the prevalence of dyspnea is now over 70%, higher than estimates reported in older cohorts. Although cancer burden, such as extensive disease in the lung or pleural effusions, certainly causes and exacerbates symptoms of breathlessness, psychological factors also underlie the experience of dyspnea. Patient-reported dyspnea is associated with impaired quality of life, decreased functioning at home and work, withdrawal from social activities, heightened symptoms of anxiety and depression, and even a desire for hastened death. Moreover, dyspnea leads to unscheduled visits to oncology clinics and the emergency department, often resulting in hospitalization. Recognizing the notable impact of breathlessness on patient functioning and health care utilization, the Quality Oncology Practice Initiative for the American Society of Clinical Oncology identified the assessment and management of dyspnea as a key measure of quality cancer care. Unfortunately, data are limited to support efficacious treatments for dyspnea. While clinicians commonly prescribe opioids to treat breathlessness, recent systematic reviews concluded that pharmacologic management did not improve dyspnea and carried potential harm. In a recent Agency for Healthcare Research and Quality Comparative Effectiveness Review of non-pharmacological interventions for dyspnea, the authors reported that behavioral and multicomponent interventions involving physical activity or rehabilitation hold the greatest promise for addressing dyspnea, despite having low strength of evidence to date. Therefore, comprehensive approaches to care incorporating behavioral interventions for dyspnea are greatly needed, given the degree of patient suffering and the lack of evidence-based protocols. To address this evidence gap, the investigators developed a brief, two-session behavioral intervention for dyspnea management in patients with advanced lung cancer called, "BREEZE." To ensure the potential for broad dissemination of BREEZE, the investigators purposefully limited the number of sessions, trained oncology nurses to serve as interventionists, and successfully transitioned to fully remote delivery during the pandemic. The investigators completed a single-center randomized controlled efficacy trial of BREEZE versus usual care in patients with advanced lung cancer and self-reported dyspnea. Patients assigned to BREEZE reported significant improvements in the primary outcome of self-reported dyspnea and functional wellbeing at week eight. However, intervention effects were not sustained by the six-month follow-up time point. The investigators now propose to build upon these encouraging findings by conducting a multi-site trial of BREEZE in a diverse patient population. Moreover, the investigators have enhanced the intervention by adding a nurse-led booster session and integrating the dyspnea management components from a digital health app that their team developed for patients with advanced lung cancer, to reinforce BREEZE's evidence-based skills and to sustain intervention effects while preserving the "low-touch" for dissemination. The investigators propose to conduct a multi-site type I hybrid effectiveness-implementation trial of BREEZE plus the booster and digital health app (i.e., BREEZE+) versus an enhanced usual care control (entailing educational resources on dyspnea management) in 420 patients with advanced lung cancer reporting dyspnea. Massachusetts General Hospital, Johns Hopkins University, and the University of Miami will serve as study sites. The nurse-led sessions and digital health app components will be available in Spanish and English to enable the recruitment of a diverse sample, and the investigators will centralize intervention delivery to facilitate implementation. Data from this study will ultimately serve as the basis for a follow-up large-scale, multi-site dissemination trial of BREEZE+.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of advanced lung cancer (i.e., non-small cell lung cancer or small cell lung cancer) or mesothelioma, not being treated with curative intent
* Self-report at least moderate dyspnea per a rating ≥4 on the validated 0-10 breathlessness item of the Edmonton Symptom Assessment Scale-Revised
* Functioning independently per an Eastern Cooperative Oncology Group Performance Status ≤2
* Ability to read and respond to questions in English or Spanish
* Receiving primary cancer care at one of the participating institutions

Exclusion Criteria:

* Significant uncontrolled psychiatric disorder or other co-morbid disease (e.g., dementia, cognitive impairment), which the treating oncology clinician reports would prohibit the patient's ability to participate in study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Patient-reported Dyspnea | 8 weeks
  To compare patient-reported dyspnea between study groups at 8 weeks using the Modified Medical Research Council Dyspnea Scale, which is a one-item self-report scale to evaluate the degree of a patient's dyspnea (score range: 0-4), with a higher score indicating worse dyspnea.

SECONDARY OUTCOMES:
Patient-reported Dyspnea-related Anxiety and Discomfort | 8 weeks
  To compare patient-reported dyspnea-related anxiety and discomfort between study groups at 8 weeks using the Cancer Dyspnea Scale, which is a 12-item self-report scale that assesses the multidimensional nature of dyspnea in patients with cancer (total scale score range: 0-48), with higher scores reflecting worse dyspnea-related effort, anxiety, and physical discomfort.
Patient-reported Physical Function | 8 weeks
  To compare patient-reported physical function between study groups at 8 weeks using the PROMIS Physical Function 8b Short Form, which is an 8-item measure that evaluates self-perceived capability of one's upper dexterity, lower extremities, and activities of daily living (total scale raw score range: 8-40), with higher scores indicating a greater level of physical function.
Patient-reported Quality of Life | 8 weeks
  To compare patient-reported quality of life between study groups at 8 weeks using the Functional Assessment of Cancer Therapy-Lung Questionnaire, which is a 36-item self-report measure of physical, social, emotional, and functional wellbeing and lung-cancer specific symptoms (total scale score range: 0-136), with higher scores indicating better overall quality of life.
Patient-reported Coping with Dyspnea | 8 Weeks
  To compare patient-reported coping with dyspnea between study groups at 8 weeks using the Chronic Respiratory Disease Questionnaire-Mastery Subscale, which is a 4-item measure assessing a patient's feeling of control and mastery over their dyspnea (score range: 1-7), with higher scores indicating greater perceived control in managing dyspnea.

OTHER OUTCOMES:
Patient-reported Dyspnea | Up to 24 weeks
  To compare average trajectories between study groups in patient-reported dyspnea across all four study time points from baseline to weeks 8, 16, and 24 using the Modified Medical Research Council Dyspnea Scale, which is a one-item self-report scale to evaluate the degree of a patient's dyspnea (score range: 0-4), with a higher score indicating worse dyspnea.
Patient-reported Dyspnea-related Anxiety and Discomfort | Up to 24 weeks
  To compare average trajectories between study groups in patient-reported dyspnea-related anxiety and discomfort across all four study time points from baseline to weeks 8, 16, and 24 using the Cancer Dyspnea Scale, which is a 12-item self-report scale that assesses the multidimensional nature of dyspnea in patients with cancer (total scale score range: 0-48), with higher scores reflecting worse dyspnea-related effort, anxiety, and physical discomfort.
Patient-reported Physical Function | Up to 24 weeks
  To compare average trajectories between study groups in patient-reported physical function across all four study time points from baseline to weeks 8, 16, and 24 using the PROMIS Physical Function 8b Short Form, which is an 8-item measure that evaluates self-perceived capability of one's upper dexterity, lower extremities, and activities of daily living (total scale raw score range: 8-40), with higher scores indicating a greater level of physical function.
Patient-reported Quality of Life | Up to 24 weeks
  To compare average trajectories between study groups in patient-reported quality of life across all four study time points from baseline to weeks 8, 16, and 24 using the Functional Assessment of Cancer Therapy-Lung Questionnaire, which is a 36-item self-report measure of physical, social, emotional, and functional wellbeing and lung-cancer specific symptoms (total scale score range: 0-136), with higher scores indicating better overall quality of life.
Patient-reported Coping with Dyspnea | Up to 24 weeks
  To compare average trajectories between study groups in patient-reported coping with dyspnea across all four study time points from baseline to weeks 8, 16, and 24 using the Chronic Respiratory Disease Questionnaire-Mastery Subscale, which is a 4-item measure assessing a patient's feeling of control and mastery over their dyspnea (score range: 1-7), with higher scores indicating greater perceived control in managing dyspnea.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Miami, Coral Gables, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The total scale, subscale scores, and item-level scores from the self-report measures, sociodemographic information, and electronic health record data will be preserved and stored within a secure computing environment. All participant identifiers will be removed and maintained in a separate secure file that will not be shared to protect confidentiality.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be submitted to a publicly available database within three months of study completion and maintained in perpetuity.
Access Criteria: Most of the scientific data generated in this study, including the self-report and electronic health record data, will be made publicly available through the Harvard Dataverse. However, certain sociodemographic information and any other variables that are considered Protected Health Information and potentially identifying the patient participants (e.g., dates of birth and death) will be restricted. Restricted data would only be made available to users who demonstrate a valid research need and meet conditions of use. In accordance with the data repository methods, we will require the completion of a data use agreement form that stipulates data sharing under IRB-approved protocols.

REFERENCES:
- [Background] Greer JA, MacDonald JJ, Vaughn J, Viscosi E, Traeger L, McDonnell T, Pirl WF, Temel JS. Pilot Study of a Brief Behavioral Intervention for Dyspnea in Patients With Advanced Lung Cancer. J Pain Symptom Manage. 2015 Dec;50(6):854-60. doi: 10.1016/j.jpainsymman.2015.06.010. Epub 2015 Jul 10. PMID 26166181
- [Background] Greer JA, Post KE, Chabria R, Aribindi S, Brennan N, Eche-Ugwu IJ, Halpenny B, Fox E, Lo S, Waldman LP, Pintro K, Rabideau DJ, Pirl WF, Cooley ME, Temel JS. Randomized Controlled Trial of a Nurse-Led Brief Behavioral Intervention for Dyspnea in Patients With Advanced Lung Cancer. J Clin Oncol. 2024 Oct 20;42(30):3570-3580. doi: 10.1200/JCO.24.00048. Epub 2024 Aug 1. PMID 39088766